CLINICAL TRIAL: NCT03903562
Title: A Phase 3 Open-Label Clinical Trial to Study the Immunogenicity and Safety of 9- Valent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) Vaccine (V503) in Chinese Females 9 to 45 Years of Age
Brief Title: Immunobridging Study of 9- Valent Human Papillomavirus (9vHPV) Vaccine (V503) in Chinese Females 9 to 45 Years of Age (V503-024)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V503-024; V503-024 (Other: MSD)
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- V503 (Experimental): V503 administered as a 0.5 mL intramuscular injection at Day 1, Month 2 and Month 6.
  Interventions: Biological: V503

INTERVENTIONS:
Biological: V503 — 0.5 mL 9vHPV VLP Vaccine

SUMMARY:
This study will investigate the immunogenicity and safety of the 9vHPV vaccine in healthy Chinese females 9 to 45 years of age. The study consists of Stage I (Day 1 to Month 7) and Stage II (post Month 7 to Month 60). Stage II will report the long-term immunogenicity and safety in the 9-19 year-old age group only. The dual-primary hypotheses of Stage I are that 9vHPV vaccine induces non-inferior immune responses in females 9 to 19 years of age who are seronegative at Day 1 to the relevant HPV type compared to females 20 to 26 years of age who are seronegative at Day 1 to the relevant HPV type, as measured by anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 GMTs at 1 month post Dose 3, and 9vHPV vaccine induces non-inferior immune responses in females 27 to 45 years of age who are seronegative at Day 1 to the relevant HPV type compared to females 20 to 26 years of age who are seronegative at Day 1 to the relevant HPV type, as measured by the seroconversion percentages to each of HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 at 1 month post Dose 3. (Each vaccine component will be analyzed separately.)

ELIGIBILITY:
Inclusion Criteria

* Participant is a Chinese female judged to be in good physical health based on medical history and physical examination
* Not a woman of childbearing potential (WOCBP) or if of WOCBP, has not had sex with males or has had sex with males and used effective contraception as defined in Appendix 2 since the first day of participant's last menstrual period through Day 1. And the participant understands and agrees that during the Day 1 through Month 7 period, she should not have sexual intercourse with males without effective contraception, and that the use of the rhythm method, withdrawal, and emergency contraception are not acceptable methods
* Has a lifetime history of 0 to 4 male and/or female sexual partners at the time of enrollment. Male partner is defined as someone with whom the participant has penile penetrative sexual intercourse. Female partner is defined as someone who has contacted, either by penetrative (with fingers or other objects) or non-penetrative means, the participant's genitalia during sexual activity

Exclusion Criteria

* Known allergy to any vaccine component, including aluminum, yeast, or BENZONASE™ (nuclease, Nycomed™). An allergy to vaccine components is defined as an allergic reaction that met the criteria for serious adverse event
* History of severe allergic reaction (e.g. swelling of the mouth and throat, difficulty breathing, hypotension, or shock) that required medical intervention
* Known thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections
* Has a fever (defined as an axillary temperature ≥37.1°C) within 24 hours prior to the Day 1 vaccination
* Has any history of abnormal Pap test showing squamous intraepithelial lesion (SIL) or atypical squamous cells - undetermined significance (ASC-US), atypical squamous cells - cannot exclude HSIL (ASC-H), atypical glandular cells, or biopsy showing cervical intraepithelial neoplasia (CIN), adenocarcinoma in situ or cervical cancer
* History of external genital wart, vulvar intraepithelial neoplasia (VIN), vaginal intraepithelial neoplasia (VaIN), vulvar cancer or vaginal cancer
* History of a positive test for HPV
* Currently immunocompromised or has been diagnosed as having congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease, or other autoimmune condition
* History of splenectomy
* Donated blood within 1 week prior to the Day 1 vaccination, or intends to donate during Day 1 through Month 7 of the study
* Expecting to donate eggs during Day 1 through Month 7 of the study
* Pregnant
* Receiving or has received in the year prior to Day 1 vaccination the following immunosuppressive therapies: radiation therapy, cyclophosphamide, azathioprine, methotrexate, any chemotherapy, cyclosporin, leflunomide (Arava™), tumor necrosis factor (TNF)-α antagonists, monoclonal antibody therapies (including rituximab [Rituxan™]), intravenous gamma globulin (IVIG), antilymphocyte sera, or other therapy known to interfere with the immune response. With regard to systemic corticosteroids, a participant will be excluded if she is currently receiving steroid therapy, has recently (defined as within 2 weeks of Day 1 vaccination) received such therapy, or has received 2 or more courses of corticosteroids (orally or parenterally) lasting at least 1 week in duration in the year prior to Day 1 vaccination. Participants using inhaled, nasal or topical corticosteroids are considered eligible for the study
* Has received immune globulin product (including RhoGAM™ or blood-derived product other than IVIG within 6 months prior to Day 1 vaccination, or plans to receive any such product during Day 1 through Month 7 of the study
* Has received a marketed HPV vaccine, or has participated in an HPV vaccine clinical trial and has received either active agent or placebo
* Has received inactivated or recombinant vaccines within 14 days prior to Day 1 vaccination or has received live vaccines within 21 days prior to Day 1 vaccination
* Concurrently enrolled in clinical studies of interventional agents
* a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence. Alcohol abusers are defined as those who drink despite recurrent social, interpersonal, and/or legal problems as a result of alcohol use

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Must be a Chinese female
Enrollment: 1990 (Actual)
Dates: Start 2019-04-27 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Stage I: Competitive Luminex Immunoassay (cLIA) GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 Years of Age and 20 to 26 Years of Age: Month 7 | 1 month post vaccination 3 (Month 7)
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type will be reported in mMU/mL.
Stage I: Percentage of Participants 27 to 45 Years of Age and 20 to 26 Years of Age Who Are Seropositive by cLIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 7 | 1 month post vaccination 3 (Month 7)
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA and will be reported in mMU/mL. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage II: cLIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 Years of Age: Month 12 | Month 12
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type will be reported in mMU/mL.
Stage II: cLIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 years of Age: Month24 | Month 24
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type will be reported in mMU/mL.
Stage II: cLIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 years of Age: Month 36 | Month 36
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type will be reported in mMU/mL.
Stage II: cLIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 years of Age: Month 48 | Month 48
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type will be reported in mMU/mL.
Stage II: cLIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 years of Age: Month 60 | Month 60
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type will be reported in mMU/mL.
Stage II: Percentage of Participants 9 to 19 Years of Age Who Are Seropositive by cLIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 12 | Month 12
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will determined using cLIA. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage II: Percentage of Participants 9 to 19 Years of Age Who Are Seropositive by cLIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 24 | Month 24
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will determined using cLIA. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage II: Percentage of Participants 9 to 19 Years of Age Who Are Seropositive by cLIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 36 | Month 36
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will determined using cLIA. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage II: Percentage of Participants 9 to 19 Years of Age Who Are Seropositive by cLIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 48 | Month 48
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will determined using cLIA. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage II: Percentage of Participants 9 to 19 years of Age Who Are Seropositive by cLIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 60 | Month 60
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will determined using cLIA. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage II: Immunoglobulin G Luminex Immunoassay (IgG LIA) GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 years of Age: Month 12 | Month 12
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The GMT for each HPV type will be reported in mMU/mL.
Stage II: IgG LIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 years of Age: Month 24 | Month 24
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The GMT for each HPV type will be reported in mMU/mL.
Stage II: IgG LIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 years of Age: Month 36 | Month 36
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The GMT for each HPV type will be reported in mMU/mL.
Stage II: IgG LIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 years of Age: Month 48 | Month 48
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The GMT for each HPV type will be reported in mMU/mL.
Stage II: IgG LIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 years of Age: Month 60 | Month 60
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The GMT for each HPV type will be reported in mMU/mL.
Stage II: Percentage of Participants 9 to 19 Years of Age Who Are Seropositive by IgG LIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 12 | Month 12
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The percentage of participants that achieve the serostatus cutoffs for seroconversion for each HPV type will be summarized.
Stage II: Percentage of Participants 9 to 19 Years of Age Who Are Seropositive by IgG LIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 24 | Month 24
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The percentage of participants that achieve the serostatus cutoffs for seroconversion for each HPV type will be summarized.
Stage II: Percentage of Participants 9 to 19 Years of Age Who Are Seropositive by IgG LIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 36 | Month 36
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The percentage of participants that achieve the serostatus cutoffs for seroconversion for each HPV type will be summarized.
Stage II: Percentage of Participants 9 to 19 Years of Age Who Are Seropositive by IgG LIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 48 | Month 48
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The percentage of participants that achieve the serostatus cutoffs for seroconversion for each HPV type will be summarized.
Stage II: Percentage of Participants 9 to 19 Years of Age Who Are Seropositive by IgG LIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 60 | Month 60
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The percentage of participants that achieve the serostatus cutoffs for seroconversion for each HPV type will be summarized.

SECONDARY OUTCOMES:
Stage I: Percentage of Participants 9 to 19 Years of Age and 20 to 26 Years of Age Who Are Seropositive by cLIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 7 | 1 month post vaccination 3 (Month 7)
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA and are reported in mMU/mL. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage I: cLIA GMTs for HPV Tys 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 15 Years of Age and 20 to 26 Years of Age: Month 7 | 1 month post vaccination 3 (Month 7)
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type will be reported in mMU/mL.
Stage I: Percentage of Participants 9 to 15 Years of Age Who Are Seropositive by cLIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 7 | 1 month post vaccination 3 (Month 7)
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA and are reported in mMU/mL. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage I: cLIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 27 to 45 Years of Age: Month 7 | 1 month post vaccination 3 (Month 7)
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type will be reported in mMU/mL.
Stage I: IgG LIA GMTs for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 in Participants 9 to 19 Years of Age, 20 to 26 Years of Age, and 27 to 45 Years of Age: Month 7 | 1 month post vaccination 3 (Month 7)
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA. The GMT for each HPV type will be reported in mMU/mL.
Stage I: Percentage of Participants 9 to 19 Years of Age, 20 to 26 Years of Age, and 27 to 45 Years of Age Who Are Seropositive by IgG LIA to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58: Month 7 | 1 month post vaccination 3 (Month 7)
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using IgG LIA and are reported in mMU/mL. The percentage of participants who are seropositive for each HPV type will be summarized.
Stage I: Percentage of Participants Who Experience at Least 1 Solicited Injection-site AE | Up to 8 days post any vaccination
  An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. The participant or the parent/guardian of the participant were to record the presence of any vaccination report card (VRC)-prompted injection-site AEs that occurred in the 8 days after any vaccination. The percentage of participants with an injection-site AE prompted on the VRC (erythema, pain, swelling and induration) will be summarized.
Stage I: Percentage of Participants Who Experience at Least 1 Systemic AE | Up to 30 days post any vaccination
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. The percentage of participants with a systemic AE will be summarized.
Stage I: Percentage of Participants Who Experience at Least 1 Serious Adverse Event (SAE) | Day 1 to Month 7
  An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the study vaccine. An SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event. The percentage of participants that experienced 1 or more SAEs will be summarized.
Stage I: Percentage of Participants with Elevated Axillary Temperature (≥37.1 C) | up to 8 days post any vaccination
  Participant or participant's legally acceptable representative will be asked to record axillary temperature in the evening after each study vaccination and daily, at the same time of day whenever possible, for 7 days after each study vaccination in the VRC. The percentage of participant's who had an axillary temperature ≥37.1°C will be summarized.
Stage II: Percentage of Participant 9 to 19 years of Age Who Experience at Least 1 Serious Adverse Event (SAE): Month 7 to Month 60 | Month 7 to Month 60
  An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the study vaccine. An SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event. The percentage of participants that experienced 1 or more SAEs will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- China (2):
  - Kaihua country Center for Disease Control and Prevention ( Site 0002), Quzhou, Zhejiang
  - Shaoxing keqiao center for disease prevention and control ( Site 0001), Shaoxing, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Lv H, Wang S, Liang Z, Yu W, Yan C, Chen Y, Hu X, Fu R, Zheng M, Group T, Luxembourg A, Liao X, Chen Z. Immunogenicity and safety of the 9-valent human papillomavirus vaccine in Chinese females 9-45 years of age: A phase 3 open-label study. Vaccine. 2022 May 20;40(23):3263-3271. doi: 10.1016/j.vaccine.2022.02.061. Epub 2022 Apr 26. PMID 35487814
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com